CLINICAL TRIAL: NCT04196920
Title: Methotrexate-associated Anti-TNF Alpha (Infliximab/Adalimumab) Combination Therapy: Evaluation of Efficacy and Safety Compared to Traditional Azathioprine-associated Combination Therapy in Patients With Chronic Inflammatory Bowel Disease.
Brief Title: Methotrexate-associated Anti-TNF Combination Therapy, the Neglected One !
Acronym: MTX
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Rennes University Hospital - CHU Pontchaillou (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0580
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Chronic Inflammatory Bowel Disease
Keywords: Crohn's disease; ulcerated ulcerative colitis
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort with TNF combination therapy: Cohort with TNF combination therapy (infiximab/adalimumab) with azathiorpine
- Cohort with anti-TNF combination therapy: Cohort with anti-TNF combination therapy (infiximab/adalimumab) with methotrexate

SUMMARY:
The results of the SONIC trial represented a significant advance in the management of patients with chronic inflammatory bowel disease by demonstrating the superiority of the combination of an alpha TNF anti-TNF with immunosuppressive therapy in naive patients (infliximab and azathioprine) compared to monotherapy in terms of clinical and endoscopic remission (40% versus 22%, p = 0.017). The benefit of this combination therapy is both pharmacological (addition, or even synergy of the two treatments) and immunological (reduction of the risk of immunization to biotherapy).

Data on the use of immunosuppressive methotrexate treatment are divergent. Indeed, a previous randomized trial suggested that the combination of anti-TNF alpha including infliximab and methotrexate was no more effective than anti-TNF alpha monotherapy in patients with Crohn's disease. However, the superiority of this combination has been clearly demonstrated over monotherapy in rheumatology for a long time.

In practice, more and more practitioners are prescribing this combination (antiTNF and MTX) in IBD patients because of tolerance problems, particularly to azathioprine or in patients with a dual expression of their disease, both digestive and joint.

The interest of my thesis work is therefore to be able to clarify these grey areas and to be able to modify or comfort therapeutic choices in practice.

DETAILED DESCRIPTION:
Data will be extracted from medical records (age, gender, smoking status, date of diagnosis of chronic inflammatory disease, date of first prescription of antiTNF alpha either infliximab or adalimumab, date of start and end of immunosuppressive azathioprine/6MP and/or metrotrexate, mode of administration of per os or SC/IV treatment, efficacy based on validated clinical scores HBI-PDAI-Mayo, tolerance). A collection will be made on the University Hospital from a computer workstation. An analysis will then be carried out to write the publication secondarily. The data retention period will be one year from November 2019 to November 2020 depending on the duration of this thesis work, which is estimated at one year.

Expected results and prospects : " Methotrexate-associated antiTNF alpha combination therapy is as effective and safe as traditional azathioprine combination therapy in patients with IBD. The positive results may in practice lead to changes in our practices and give first priority to this combination therapy with methotrexate. "

ELIGIBILITY:
Inclusion criteria :

- Patients with chronic inflammatory bowel disease including Crohn's disease and ulcerated rectocolitis under combination therapy with anti-TNF alpha

Exclusion criteria:

Subject unable to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic inflammatory bowel disease including Crohn's disease and ulcerated rectocolitis under combination therapy with anti-TNF alpha (infliximab, adalimumab) from January 2013 to November 2019
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of anti-TNF alpha and methotrexate combination therapy | through study completion, an average of 7 years
  Evaluation of the efficacy of anti-TNF alpha and methotrexate combination therapy compared to conventional azathioprine combination therapy. Efficacy is defined according to response and remission without corticosteroids based on clinical scores, biological markers, endoscopic criteria and immunization rates.

SECONDARY OUTCOMES:
Tolerance assessment of anti-TNF alpha and methotrexate combination therapy | 6 months, one year, two years, and date on the latest news
  Tolerance assessment of anti-TNF alpha and methotrexate combination therapy compared to conventional azathioprine combination therapy. Number of stops for treatment intolerance, minor adverse events, severe adverse events, infection rate, cancer risk

CONTACTS AND LOCATIONS:
Overall Officials: Najima BOUTA, Resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC